CLINICAL TRIAL: NCT00033644
Title: A Phase II Evaluation of DMAP Plus GM-CSF in the Treatment of Advanced, Persistent, or Recurrent Leiomyosarcoma of the Uterus
Brief Title: Combination Chemotherapy Plus Sargramostim in Treating Patients With Cancer of the Uterus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000069308; GOG-0087K
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2004-09

CONDITIONS: Sarcoma
Keywords: stage IV uterine sarcoma; recurrent uterine sarcoma; uterine leiomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — sargramostim; Cisplatin; Dacarbazine; Doxorubicin; Mitomycin

INTERVENTIONS:
Biological: sargramostim
Drug: cisplatin
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: mitomycin C

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus sargramostim in treating patients who have advanced, persistent, or recurrent cancer of the uterus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of dacarbazine, mitomycin, doxorubicin, and cisplatin plus sargramostim (GM-CSF) in patients with advanced, persistent, or recurrent leiomyosarcoma of the uterus.
* Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE: Patients receive dacarbazine IV over 2 hours, followed by mitomycin IV over 2-5 minutes, doxorubicin IV over 2-5 minutes, and cisplatin IV over 2 hours on day 1. Patients also receive sargramostim (GM-CSF) subcutaneously (SC) once every 12 hours on days -6 to -3 before the first chemotherapy course and then on days 2-15 and 23-26 of all chemotherapy courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease receive a maximum of 4 courses. Patients achieving complete or partial response receive a maximum of 6 courses.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 12-43 patients will be accrued for this study within 12-28 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary leiomyosarcoma (LMS) of the uterus

  * Advanced, persistent, or recurrent disease that is refractory to curative therapy or established treatments
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques (e.g., palpation, plain x-ray, CT scan, or MRI) OR
  * At least 10 mm by spiral CT scan
  * Tumors within a previously irradiated field are designated as non-target lesions
* Ineligible for a higher priority Gynecologic Oncology Group protocol (if one exists), including any active phase III protocol for the same population

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* No active infection requiring antibiotics
* No grade 2 or greater sensory or motor neuropathy
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior cytotoxic chemotherapy for LMS of the uterus

Endocrine therapy:

* At least 1 week since prior hormonal therapy for LMS of the uterus
* Concurrent hormone replacement therapy allowed

Radiotherapy:

* See Disease Characteristics
* Recovered from prior recent radiotherapy

Surgery:

* Recovered from prior recent surgery

Other:

* Recovered from other prior recent therapy
* No prior cancer treatment that would preclude study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03; Primary Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry J. Long, MD, Study Chair — Mayo Clinic
Locations (21):
- United States (20):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Tuft-New England Medical Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, Cincinnati, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Tacoma General Hospital, Tacoma, Washington
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Long HJ 3rd, Blessing JA, Sorosky J. Phase II trial of dacarbazine, mitomycin, doxorubicin, and cisplatin with sargramostim in uterine leiomyosarcoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2005 Nov;99(2):339-42. doi: 10.1016/j.ygyno.2005.06.002. Epub 2005 Jul 26. PMID 16051328